CLINICAL TRIAL: NCT05802667
Title: A Cohort Study of Correlation Between Mast Cells and Prognosis in Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2023124
Record Dates: First submitted 2023-03-26; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Inflammation; Acute ST Segment Elevation Myocardial Infarction; Prognosis
MeSH Terms: conditions — Inflammation; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples were collected from patients within 24 hours, 1 month, 3 months and 12 months after myocardial infarction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI: A total of 300 STEMI patients admitted to the Department of Cardiology, Peking University Third Hospital from April 1, 2023 to March 31, 2024 were enrolled.
  Interventions: Diagnostic Test: Tryptase

INTERVENTIONS:
Diagnostic Test: Tryptase — Serum samples were collected from patients within 24 hours, 1 month, 3 months and 12 months after myocardial infarction, and trypsin-like enzymes were determined by elisa

SUMMARY:
By including patients with acute myocardial infarction, mast cell markers were analyzed and the relationship between mast cells and patients with acute myocardial infarction was analyzed

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is the best way to improve the prognosis of patients with acute ST-segment elevation myocardial infarction (STEMI). However, ischemia reperfusion injury, inappropriate ventricular remodeling, and myocardial fibrosis may still be present in STEMI after PCI, which may be related to the inflammatory response in STEMI. Mast cells (MC), their degranulation products and induction of a series of inflammatory cytokines play an important role in the inflammatory response. The purpose of this study was to evaluate the relationship between mast cell markers (trypsin, chymotrypsin) levels and prognosis after direct PCI in STEMI patients. We prospectively and continuously included STEMI patients undergoing standard therapy after direct PCI. Clinical data and blood samples were collected and followed up for 1 year to analyze mast cell markers and myocardial infarction size. As well as differences in echocardiography, markers of two-dimensional speck tracking techniques, inflammatory factors and major adverse cardiovascular events, to explore the relationship between mast cells and their products and ventricular remodeling and ischemia-reperfusion injury in STEMI patients, and to provide new ideas for treatment and new basis for optimization of STEMI treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old, regardless of gender;
* 2) Meet STEMI diagnostic criteria (diagnostic criteria: ischemic chest pain lasting ≥30min; ST segment elevation of more than two adjacent leads or new left bundle branch block in ECG; With or without elevated myocardial markers) and receiving standard care for STEMI.
* 3) Agree to and cooperate with the study

Exclusion Criteria:

* 1) The patient is taking or planning to take long-term oral or intravenous glucocorticoids (inhaled and topical hormones are allowed);
* 2) Allergic diseases, autoimmune diseases or malignant tumors.
* 3) Patients with metal implants or claustrophobia are not allowed to undergo an MRI examination;
* 4) Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three hundred STEMI patients who meet the inclusion criteria and do not meet the exclusion criteria admitted to the Department of Cardiovascular Medicine of Peking University Third Hospital were continuously recruited.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size | 3 months after myocardial infarction
  Myocardial infarct size was assessed by cardiac MRI

SECONDARY OUTCOMES:
left ventricular systolic function | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
  Transthoracic echocardiography to measure LVEF, left ventricular end-diastolic diameter, Em/Sm
Left ventricular ultrasound strain | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
  Two-dimensional speckle tracking imaging measures the movement in the long-axis direction as the overall longitudinal strain, the movement in the short-axis direction as the overall radial strain, reflecting the degree of wall systolic thickening, and the annular motion in the short-axis direction as the overall circumferential strain
inflammatory marker such as TNF-α | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
inflammatory markers e.g. IL1, IL6 | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
MC marker (chymotrypsin) | 24 hours, 1 month, 3 months, and 12 months after myocardial infarction
major adverse cardiovascular events | 12 months
  MACE events (death, nonfatal myocardial infarction, unplanned revascularization, hospitalization for angina and readmission for heart failure)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Cui, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie P, Xu S, Chen X, Xu H, Zhang R, Li D, Sun L, Zhu D, Cui M. Tryptase as a Biomarker for Adverse Prognosis in ST-Segment Elevation Myocardial Infarction Patients: A Prospective Cohort Study. J Inflamm Res. 2025 Mar 14;18:3817-3828. doi: 10.2147/JIR.S502496. eCollection 2025. PMID 40103802